CLINICAL TRIAL: NCT06068478
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial, Efficacy and Safety Study of Qingzhu Granules in the Treatment of Acute Gouty Arthritis ( Damp Heat Pattern)
Brief Title: A Study to Evaluate Efficacy and Safety of Qingzhu Granules in the Treatment of Acute Gouty Arthritis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-QZKL-Ⅲ
Record Dates: First submitted 2023-09-27; First posted 2023-10-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-10

CONDITIONS: Gouty Arthritis
MeSH Terms: conditions — Arthritis, Gouty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qingzhu Granules (Experimental)
  Interventions: Drug: Qingzhu Granules
- Qingzhu Granules Placebo (Placebo Comparator)
  Interventions: Drug: Qingzhu Granules Placebo

INTERVENTIONS:
Drug: Qingzhu Granules — During the 72-hour treatment period, participants will receive 9 sacks of Qingzhu granules.Oral administration, 1 sack (6g) per time, 3 times daily.
  Arms: Qingzhu Granules
Drug: Qingzhu Granules Placebo — During the 72-hour treatment period, participants will receive 9 sacks of Qingzhu granules Placebo.Oral administration, 1 sack (6g) per time, 3 times daily.
  Arms: Qingzhu Granules Placebo

SUMMARY:
This study will evaluate the efficacy and safety of Qingzhu Granules in the treatment of Acute Gouty Arthritis ( Damp heat pattern)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 to 70 years.
2. Patient meeting the ACR/ EULAR 2015 gout classification criteria.
3. Patient meeting the Damp heat Pattern identification of the traditional Chinese medicine.
4. Onset of current flare within 48 hours.
5. Patient-reported, current ongoing flare of gouty arthritis characterized by baseline pain intensity in the index joint of ≥40 mm on a 0-100 mm VAS.
6. Signed informed consent to participate in this study.

Exclusion Criteria:

1. Secondary gouty arthritis ( caused by other diseases or drugs).
2. The presence of pain symptoms caused by other diseases, as judged by the investigator, may have an impact on the safety or effectiveness evaluation.
3. If there are severe motor, digestive, respiratory, urological, reproductive, endocrine, immune, neurological, circulatory, or psychiatric disorders, the investigator may determine that it may have an impact on the safety or effectiveness evaluation.
4. Abnormal liver function (glutamic-oxaloacetic transaminase or glutamic-pyruvic transaminase>2 ULN) or abnormal renal function (blood creatinine>ULN).
5. People who are not eligible for VAS evaluation, such as those with severe impairment of abstract ability, visual and writing function, and those who have taken sedatives.
6. Patients who have undergone uric acid lowering treatment but have not stably used uric acid lowering drugs within the 2 weeks prior to randomization.
7. After this gout attack, traditional Chinese medicine, chemical drugs (including but not limited to colchicine, glucocorticoids, and adrenocorticotropins), biological drugs (including but not limited to IL-1 and TNF- α Inhibitor) ,and non drug treatment (including but not limited to acupuncture and moxibustion and topical ice)that have therapeutic effects on gout have been used.
8. After this gout attack, non-steroidal anti-inflammatory drugs (including but not limited to aspirin, acetaminophen, losoprofen, ibuprofen, and diclofenac sodium) have been used, and the medication duration is within 5 half-lives of the drug.
9. Known allergies to the drug components of this study.
10. Contraindications to diclofenac sodium enteric coated tablets.
11. Men or women who have plans for conception within 3 months after the start to the end of the study.
12. Pregnant and lactating women.
13. Participated in other clinical trials within the past month.
14. Other situations that the investigator determines are not suitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | 72 hours
  Change from basline in Patient-assessed Pain Intensity on VAS at 72 hours after the investigational product therapy.

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) | 24/48 hours
  Change from basline in Patient-assessed Pain Intensity on VAS at 24/48 hours.
The total score of the Traditional Chinese Medicine Syndrome | 72 hours
  Change from basline in the total score of the Traditional Chinese Medicine Syndrome Scoring Scale at 72 hours.
The each item score of the Traditional Chinese Medicine Syndrome | 72 hours
  Change from basline in each item of the Traditional Chinese Medicine Syndrome Scoring Scale at 72 hours.
CRP | 72 hours
  Change from baseline in the inflammatory biomarkers CRP and at 72 hours.
Rescue medication | 72 hours
  The total dose and frequency of rescue medication use within 72 hours of treatment.
Time interval | 72 hours
  The interval between the first use of emergency medication and the first use of Investigational Product.

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Henan Province Luoyang Orthopedic Hospital, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Guang'anmen Hospital of the Chinese Academy of Traditional Chinese Medicine, Beijing
  - Binzhou Medical College Affiliated Hospital, Binzhou
  - Bozhou People's Hospital, Bozhou
  - Hebei Cangzhou Integrated Traditional Chinese and Western Medicine Hospital, Cangzhou
  - The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine, Changsha
  - Dalian Central Hospital, Dalian
  - The First Affiliated Hospital of Hainan Medical College, Haikou
  - Hebei Provincial People's Hospital, Hebei
  - The First Affiliated Hospital of South China University, Hengyang
  - Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan
  - The First Affiliated Hospital of Kunming Medical University, Kunming
  - Yunnan First People's Hospital, Kunming
  - Yunnan Provincial Traditional Chinese Medicine Hospital, Kunming
  - Gansu Provincial Hospital of Traditional Chinese Medicine, Lanzhou
  - Gansu Provincial People's Hospital, Lanzhou
  - Ma'anshan People's Hospital, Ma’anshan
  - Mianyang Central Hospital, Mianyang
  - Mianyang Traditional Chinese Medicine Hospital, Mianyang
  - Pu'er People's Hospital, Pu'er
  - Puyang Oilfield General Hospital, Pujiang
  - Puyang People's Hospital, Pujiang
  - Shiyan City People's Hospital, Shiyan
  - Wenzhou People's Hospital, Wenzhou
  - Xi'an Daxing Hospital, Xi'an
  - Xiamen Traditional Chinese Medicine Hospital, Xiamen
  - Zhengzhou People's Hospital, Zhengzhou
  - Hunan Province Directly Affiliated TCM Hospital, Zhuzhou